CLINICAL TRIAL: NCT05539339
Title: Molecular Profiling of Tumor in Situ Fluid in Guiding Individualized Treatment Plan in Adults With ctDNA-level-relapse Glioblastoma
Brief Title: Personalized Trial in ctDNA-level-relapse Glioblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPPH-ttrGBM
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Open-label, pilot, umbrella trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): This arm includes patients with ctDNA-level-relapse glioblastoma before imaging recurrence.
  Interventions: Other: Individualized intervention based on genomic alterations

INTERVENTIONS:
Other: Individualized intervention based on genomic alterations — Specialized tumor board recommended agents that target the specific recurrence-driving genomic alterations that are determined by serial TISF ctDNA analysis.

SUMMARY:
Tumor in situ fluid (TISF) refers to the fluid within the surgical cavity of patients with glioblastoma. Postoperative serial TISF is collected for circulating tumor DNA (ctDNA) analysis and identifying ctDNA-level relapse driven by one or a set of specific genomic alterations before overt imaging recurrence of the tumor. This single-arm open-label prospective pilot feasibility trial recruiting 20 adult patients with ctDNA-level-relapse glioblastoma who are assigned to receive the personalized study treatment based on the genetic profile of their serial TISF ctDNA. It will be aimed to test whether the personalized intervention can prolong the progression-free and overall survival and the feasibility of conducting a full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study, including disease assessment by MRI and tumor in situ fluid (TISF) collection
3. Histologically confirmed diagnosis of glioblastoma
4. Resection surgery done at the study center (Henan Provincial People's Hospital), with a reservoir intraoperatively implanted connecting the surgical cavity and the subscalp for postoperative noninvasive TISF collection
5. Previous first line treatment with at least radiotherapy
6. An interval of > 28 days and full recovery (i.e., no ongoing safety issues) from surgical resection prior to grouping
7. Karnofsky performance status (KPS) of 70 or higher
8. Life expectancy > 12 weeks

Exclusion Criteria:

1. More than two recurrences of GBM
2. Presence of extracranial metastatic, significant leptomeningeal disease or tumors primarily localized to the brainstem or spinal cord
3. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
4. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring chronic and systemic immunosuppressive treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects have any other condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 14 days. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalent are permitted in absence of active autoimmune disease
5. Previous radiation therapy with anything other than standard radiation therapy (i.e., focally directed radiation) administered as first line therapy
6. Previous treatment with carmustine wafer except when administered as first line treatment and at least 6 months prior to randomization
7. Previous bevacizumab or other VEGF or anti-angiogenic treatment
8. Previous treatment with a PD-1, PD-L1 or CTLA-4 targeted therapy
9. Evidence of > Grade 1 CNS hemorrhage on the baseline MRI scan
10. Inadequately controlled hypertension (defined as systolic blood pressure ≥160 mmHg and /or diastolic blood pressure ≥100 mmHg) within 7 days of first study treatment
11. Prior history of hypertensive crisis, hypertensive encephalopathy, reversible posterior leukoencephalopathy syndrome (RPLS)
12. Prior history of gastrointestinal diverticulitis, perforation, or abscess
13. Clinically significant (i.e., active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
14. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment. Any previous venous thromboembolism ≥ NCI CTCAE Grade 3 within 3 months prior to start of study treatment
15. History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month prior to randomization
16. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
17. Current or recent (within 10 days of study enrollment) use of anticoagulants that, in the opinion of the investigator, would place the subject at significant risk for bleeding. Prophylactic use of anticoagulants is allowed
18. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study
19. Minor surgical procedure (e.g., stereotactic biopsy within 7 days of first study treatment; placement of a vascular access device within 2 days of first study treatment)
20. History of intracranial abscess within 6 months prior to randomization;
21. History of active gastrointestinal bleeding within 6 months prior to randomization
22. Serious, non-healing wound, active ulcer, or untreated bone fracture
23. Subjects unable (due to existent medical condition, e.g., pacemaker or ICD device) or unwilling to have a head contrast enhanced MRI
24. Positive test for hepatitis B virus surface antigen (HBV sAg) or detectable hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection
25. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
26. History of severe hypersensitivity reaction to any monoclonal antibody
27. Patients that require decadron > 4 mg/ day or equivalent of steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | Up to six months after beginning treatment
  The proportion of participants in the analysis population who remain progression-free for at least six months following initiation of study therapy.
Overall survival rate at 18 months | Up to 18 months after beginning therapy
  OS-18 is the proportion of participants in the analysis population who remain alive for at least twelve months following initiation of study therapy.

SECONDARY OUTCOMES:
Overall survival | Up to 3 years after beginning treatment
  overall survival, as defined as time from beginning of treatment to death.
Progression-free survival | Up to 3 years after beginning treatment
  Median time from allocation to first documented disease progression as per the response assessment in neuro-oncology criteria or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Xingyao Bu, MD, PhD, Study Director — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No